CLINICAL TRIAL: NCT03441282
Title: Precision Medicine in Anesthesia: Genetic Component in Opioid-induced Respiratory Depression
Status: Terminated | Type: Observational
Why Stopped: Investigator decision
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Kevin Harrod, Primary Investigator, University of Alabama at Birmingham
Other Study IDs: F23456789; UAB (Other: Anesthesiology)
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Depression
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Fentanyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ASA Patients I: Age 18-80 years old, English-speaking, not on current Fentanyl/opioid therapy, no use of opioid medications in the 3 months prior to surgery, scheduled for elective surgery at UAB main.
  A normal healthy patient Healthy, non-smoking, no or minimal alcohol use
  Interventions: Drug: Fentanyl
- ASA Patients III: Age 18-80 years old, English-speaking, not on current Fentanyl/opioid therapy, no use of opioid medications in the 3 months prior to surgery, scheduled for elective surgery at UAB main.
  A patient with severe systemic disease Substantive functional limitations; One or more moderate to severe diseases. Examples include (but not limited to): poorly controlled DM or HTN, COPD, morbid obesity (BMI ≥40), active hepatitis, alcohol dependence or abuse, implanted pacemaker, moderate reduction of ejection fraction, ESRD undergoing regularly scheduled dialysis, premature infant PCA < 60 weeks, history (>3 months) of MI, CVA, TIA, or CAD/stents.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — After the patient is attached to an ASA non-invasive monitor, a dose (2mcg/kg) of Fentanyl will be administered.
  Groups compared would include patients experiencing respiratory depression vs those not experiencing respiratory depression after fentanyl administration. Their samples would be evaluated for any differences in genetic make-up concerning selected, known sequences affecting opioid-induced analgesia.
  Other Names: Denpax; Durogesic

SUMMARY:
The concept of precision medicine - taking individual variability into account when planning preventions and interventions - is not new but is quickly gaining attention in this age of powerful methodology of patient characterization and development of tools to analyze large sets of data. Oncology is the most obvious field in which this information has been readily applied. Increasing focus, nationally and internationally, on developing broad databases of patient genetic information and research efforts evaluating those data will, hopefully, lead to the development and application of evidence-based data enhancing the practice of all fields of medicine. It has yet to become obvious how this information can best be applied to the field of anesthesiology. Most genomics work in anesthesia has been focused in the area of pain medicine. There is a known genetic influence on the potency of opioid-induced analgesia, however; a genetic component of opioid-induced respiratory depression has yet to be thoroughly evaluated. Respiratory depression plays a role in clinical care - from procedures requiring sedation with monitored anesthesia care to treating post-opertative pain and chronic pain - but perhaps its largest current role in the public arena is the unfortunate deaths caused by side effects due to drug overdose.

Personalized medicine remains on the horizon for the field of anesthesia, but, as genetic testing becomes more affordable and mainstream in clinical practice, the potential applications are broad. Most readily would be its incorporation into development of patient specific pain regimens. Respiratory depression is a potentially lethal side effect of opioid therapy. In light of the opioid epidemic and CDC-scrutiny of opioid use, determining genetic profiles susceptible to respiratory depression could prove useful in further tailoring the treatment of pain both in the perioperative setting and in the chronic pain management setting.

DETAILED DESCRIPTION:
This would be a prospective study for which patients not prescribed chronic pain medication (defined as not using narcotic medications in 3 months prior to surgery) and presenting for surgery would be recruited. Preop administration of sedating medications (i.e. midazolam) would be avoided. On the day of surgery, once in OR and standard ASA monitors placed, a standardized dose of 2mcg/kg ideal body weight IV fentanyl is administered. The patient is then monitored for respiratory depression for 5 minutes prior to administration of additional induction agents. [would include respiratory rate, with RR < 10, or O2 Sat < 90%]. Would not provide supplemental oxygen during this time unless patient was already on supplemental oxygen. Patient would then be preoxygenated and general anesthesia induced. Once general anesthesia is induced, a blood sample is collected and stored. [sample could also be collected in preop upon IV placement]. Blood will be tested for Single Nucleotide Polymorphisms of genes related to opioid-induced analgesia. [Potential target genes listed in 7.0-1] This genomic data will be evaluated for any correlations of the presence of opioid-related SNPs and concomitant opioid-induced respiratory depression.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old,
* English-speaking,
* Not on current opioid therapy,
* ASA I-III,
* Scheduled for elective surgery at UAB main

Exclusion Criteria:

* Chronic opioid therapy [Consistent use of opioid meds 3 months prior to surgery]
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from the OR schedule and recruit/consent patients in the preop clinic or preop holding area during preop evaluation.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Single Nucleotide Polymorphisms | 5 min Preop
  Preop-Blood will be tested for Single Nucleotide Polymorphisms of genes related to opioid-induced analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Tim Ness, MD, PhD, Study Chair — UAB Anesthesiology and Perioperative Medicine
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided